CLINICAL TRIAL: NCT07372976
Title: The Role and Outcome of Upper Gastrointestinal Endoscopy in Children Presenting With Chronic Abdominal Pain at Assiut University Children Hospital
Brief Title: Role and Diagnostic Yield of Upper Endoscopy in Children With Chronic Abdominal Pain
Acronym: UGI-CAP
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Randa Mahmoud Amin Mahran, Randa Mahmoud Amin Mahran, Assiut University
Other Study IDs: AUC-PED-GI-CAP-2026
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Gastrointestinal Disorders; Chronic Abdominal Pain in Children
Keywords: Chronic abdominal pain; Paediatric abdominal pain; Functional abdominal pain; Organic gastrointestinal disease; Children; Alarm symptoms; Upper gastrointestinal endoscopy; Paediatric gastroenterology; Esophagogastroduodenoscopy
MeSH Terms: interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biopsy specimens are obtained for histopathological diagnosis only, with no genetic or DNA analysis planned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with chronic abdominal pain: This group includes children aged 18 years or younger presenting with chronic abdominal pain lasting at least three months who undergo upper gastrointestinal endoscopy as part of their routine clinical evaluation at Assiut University Children Hospital. Clinical features, alarm symptoms, endoscopic findings, and histopathological results will be analyzed.
  Interventions: Diagnostic Test: Upper Gastrointestinal Endoscopy

INTERVENTIONS:
Diagnostic Test: Upper Gastrointestinal Endoscopy — Upper gastrointestinal endoscopy (esophagogastroduodenoscopy) is performed as part of standard clinical care to evaluate children with chronic abdominal pain. The procedure allows direct visualization of the esophagus, stomach, and duodenum, with biopsy sampling when clinically indicated for histopathological examination. The procedure is not assigned by the study protocol but is analyzed observationally.

SUMMARY:
Chronic abdominal pain is a common problem in children and may be caused by functional or organic gastrointestinal disorders. While many children have no identifiable structural disease, some may have conditions that can be detected by upper gastrointestinal endoscopy. This study aims to evaluate the role and diagnostic outcome of upper gastrointestinal endoscopy in children presenting with chronic abdominal pain at Assiut University Children Hospital.

Children aged 18 years or younger who have had abdominal pain for at least three months and who undergo upper gastrointestinal endoscopy as part of their routine medical care will be included. Clinical symptoms, alarm features, endoscopic findings, and biopsy results will be analyzed to determine how often endoscopy identifies an organic cause of pain. The results of this study may help guide the appropriate use of endoscopy in the evaluation of chronic abdominal pain in children.

DETAILED DESCRIPTION:
Chronic abdominal pain in children represents a frequent and challenging clinical problem. Although the majority of affected children suffer from functional gastrointestinal disorders, a significant proportion may have underlying organic diseases such as gastritis, gastroesophageal reflux disease, peptic ulcer disease, celiac disease, or other inflammatory conditions. Differentiating between functional and organic causes is essential to guide appropriate management and avoid unnecessary investigations.

Upper gastrointestinal endoscopy allows direct visualization of the esophagus, stomach, and duodenum, as well as the ability to obtain tissue biopsies for histopathological evaluation. Despite its diagnostic potential, the routine use of endoscopy in children with chronic abdominal pain remains controversial, particularly in the absence of alarm symptoms. Current guidelines suggest that endoscopy should be reserved for selected patients, but data on its diagnostic yield in pediatric populations remain limited.

This analytic cross-sectional observational study will be conducted at the Pediatric Gastroenterology and Hepatology Unit of Assiut University Children Hospital over a one-year period from January 2026 to December 2026. The study will include children aged 18 years or younger who present with chronic abdominal pain lasting at least three months and who undergo upper gastrointestinal endoscopy as part of their clinical evaluation.

All enrolled patients will undergo detailed clinical assessment, including medical history, evaluation of abdominal pain characteristics, presence of dyspeptic symptoms, and identification of alarm features such as weight loss, poor growth, gastrointestinal bleeding, persistent vomiting, chronic diarrhea, unexplained fever, abdominal mass, or organomegaly. Pain severity will be assessed using a standardized pain scoring scale. Physical examination findings and relevant laboratory investigations performed prior to endoscopy will be recorded.

Upper gastrointestinal endoscopy findings, including esophageal, gastric, and duodenal abnormalities, will be documented. Biopsy specimens obtained during the procedure will be examined histopathologically, and the results will be correlated with clinical and endoscopic findings. The primary outcome of the study is the diagnostic yield of upper gastrointestinal endoscopy, defined as the proportion of patients with abnormal endoscopic and/or histopathological findings. Secondary outcomes include the pattern of endoscopic diagnoses and the association between alarm features and abnormal findings.

Data will be analyzed using appropriate statistical methods to describe clinical characteristics and outcomes. The findings of this study are expected to provide valuable insight into the usefulness of upper gastrointestinal endoscopy in children with chronic abdominal pain and may help refine clinical decision-making regarding its appropriate use in pediatric practice.

ELIGIBILITY:
Inclusion Criteria:

* Children aged ≤18 years.
* Suffering from chronic abdominal pain lasting ≥3 months.
* Undergoing upper gastrointestinal endoscopy at Assiut University Children Hospital.

Exclusion Criteria:

* Pre-existing chronic diseases that may alter symptoms, such as inflammatory bowel disease or liver disease (unless these are diagnosed as a result of the study).
* Patients with "alarm symptoms" that require urgent, immediate intervention, such as active gastrointestinal bleeding.
* Patients or guardians who refuse to participate.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population consists of pediatric patients (up to 18 years old) presenting to the pediatric gastroenterology and hepatology unit of Assiut University Children Hospital with a primary complaint of chronic abdominal pain lasting at least 3 months. The estimated sample size is approximately 130 pediatric patients.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield of Upper Gastrointestinal Endoscopy | At the time of upper gastrointestinal endoscopy during the study period (January 2026-December 2026)
  Diagnostic yield is defined as the proportion of children with chronic abdominal pain who have abnormal findings detected by upper gastrointestinal endoscopy and/or histopathological examination of biopsy specimens.

SECONDARY OUTCOMES:
Pattern of Endoscopic and Histopathological Findings | At the time of upper gastrointestinal endoscopy during the study period (January 2026-December 2026)
  Assessment of the types and frequencies of abnormal endoscopic findings (esophageal, gastric, and duodenal) and corresponding histopathological diagnoses among children with chronic abdominal pain.
Association Between Alarm Features and Abnormal Endoscopic Findings | At the time of upper gastrointestinal endoscopy during the study period (January 2026-December 2026)
  Evaluation of the relationship between the presence of alarm symptoms (such as weight loss, gastrointestinal bleeding, persistent vomiting, poor growth, or chronic diarrhea) and abnormal upper gastrointestinal endoscopic or histopathological findings.
Severity of Abdominal Pain in Relation to Endoscopic Findings | At the time of clinical assessment and upper gastrointestinal endoscopy during the study period (January 2026-December 2026)
  Correlation between abdominal pain severity assessed using a standardized pain score and the presence or absence of abnormal endoscopic or histopathological findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adeniyi OF, et al. Recurrent abdominal pain and upper gastrointestinal endoscopy findings in children and adolescents. PLoS One. 2019;14(5).
- [Background] Thakkar K, Dorsey F, Gilger MA. Impact of Endoscopy on Management of Chronic Abdominal Pain in Children. Dig Dis Sci. 2010;56(2):488-493.
- [Background] Wani MA, et al. Endoscopic Yield, Appropriateness, and Complications of Pediatric Upper Gastrointestinal Endoscopy in an Adult Suite. Clin Endosc. 2020;53(4):436-442.
- [Background] Vakil N, et al. The Montreal definition and classification of gastroesophageal reflux disease. Am J Gastroenterol. 2006;101(8).
- [Background] Oka P, et al. Global prevalence of irritable bowel syndrome according to Rome III or IV criteria. Lancet Gastroenterol Hepatol. 2020;5(10):908-917.
- [Background] Berger MY, Gieteling MJ, Benninga MA. Chronic abdominal pain in children. BMJ. 2007;334(7601):997-1002. doi:10.1136/BMJ.39189.465718.BE